CLINICAL TRIAL: NCT01772264
Title: An Investigator And Subject Blinded, Sponsor Open, Randomized, Placebo Controlled, Multiple Dose Study To Investigate The Safety, Toleration And Pharmacokinetics Of Multiple Oral Doses Of PF-05089771 In Healthy Subjects
Brief Title: Safety And Tolerability Study Of BID Titration Scheme With PF-05089771
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B3291018
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
MeSH Terms: interventions — PF-05089771

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A - active treatment (Experimental)
  Interventions: Drug: PF-05089771
- Arm B - placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-05089771 — titration from 150mg BID to 450mg BID
  Arms: Arm A - active treatment
Drug: Placebo — matched placebo
  Arms: Arm B - placebo

SUMMARY:
The most notable tolerability finding from these multiple dosing studies has been the occurrence of mild to moderate rash at doses of 450 mg BID and 600 mg BID. Based upon this finding, the current four week study is designed to examine whether a slow titration regimen up to a lower maintenance dose of 450 mg BID is able to reduce the incidence of rash.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-child bearing potential between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal (ie, recurrent nephrolitisis), endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* History of, or presence of allergic skin reactions or active skin disease (except for subjects with acne who may be included in the study) at the time of screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Treatment-Related Adverse Events (AEs) or Serious Adverse Events (SAEs) | 28 days
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | 12h
Maximum Observed Plasma Concentration (Cmax) | 12h

SECONDARY OUTCOMES:
Minimum Observed Plasma Trough Concentration (Cmin) | 12h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3291018&StudyName=Safety%20And%20Tolerability%20Study%20Of%20BID%20Titration%20Scheme%20With%20PF-05089771